CLINICAL TRIAL: NCT03304860
Title: Child-Physician Recommendation on Parental Adherence to Colorectal Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 17-00570
Record Dates: First submitted 2017-10-04; First posted 2017-10-09 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CRC screening Survey (Experimental): Residents with parents eligible for CRC screening will be asked to provide their e-mail address, solely for the use of distributing the follow up survey so it can be linked to 2 brief (3-5 min) surveys
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Survey with 4-7 questions about each parents' demographics and CRC screening history. Depending on answers, provided a CRC screening document and asked to discuss screening with parents, followed by a brief survey in 4 months

SUMMARY:
Physician recommendation has been shown to be one of the most significant predictors for colorectal cancer (CRC) screening. This study aims to identify the amount of parents of internal medicine residents at NYU who are eligible for CRC screening but have not received it. Investigators will perform an intervention and quantify the amount of parents eligible for CRC screening after the intervention. This study will entail sending 2 brief surveys (one before the intervention and one after) which determine if the parents of the residents are eligible for CRC screening. The intervention will be asking the residents with eligible parents to have a discussion with their parents about CRC screening options and to address their concerns. Investigators will provide a one page document the residents can give their parents as a reference as part of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Internal medicine residents at NYU - PGY1, PGY2, and PGY3 during 2017-2018 academic year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Change in CRC screening rate of eligible parents of internal medicine residents at NYU from before to after the intervention | Baseline to 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pochapin, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No